CLINICAL TRIAL: NCT03325465
Title: Neoadjuvant Pembrolizumab + Epacadostat Prior to Curative Surgical Care for Squamous Cell Carcinoma of the Head and Neck (SCCHN): The KEO Trial
Brief Title: Neoadjuvant Pembrolizumab + Epacadostat Prior to Curative Surgical Care for Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Site decided not to move forward with trial. Study never opened to enrollment.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0993
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: squamous cell carcinoma of the head and neck; head and neck cancer; neoadjuvant pembrolizumab; epacadostat
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and epacadostat (Experimental): Patients will receive neoadjuvant immunotherapy either with anti-PD-1 (pembrolizumab) alone or anti-PD-1 in combination with IDO1 inhibition (epacadostat). Patients will receive Pembrolizumab every 3 weeks over a period of 8 weeks as well as epacadostat starting on day 1 for the duration of pembrolizumab treatment.
  All patients will undergo baseline biopsy (mandatory, sampling ≥ 4 areas to represent the tumor), as well as baseline imaging (and for exploratory analysis collection of blood for baseline ctDNA testing and TCR analysis).
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Patients will receive pembrolizumab alone or pembrolizumab in combination with epacadostat. Pembrolizumab will be administered at 200 mg IV every 3 weeks for up to 3 doses for no longer than 8 weeks prior to surgery. After surgery, patients will continue pembrolizumab plus epacadostat every 3 weeks for 12 months.
  Other Names: Keytruda
Drug: Epacadostat — Patients will receive epacadostat in combination with pembrolizumab. Epacadostat will be administered orally at a dose of 100 mg twice a day starting on day 1 for the duration of pembrolizumab treatment. Patients will continue on this combination for no longer than 8 weeks prior to surgery. After surgery, patients will continue pembrolizumab plus epacadostat every 3 weeks for 12 months.

SUMMARY:
The KEO study is a single arm phase II trial including 44 patients with T1N1-2B, T2N0-N2B head and neck squamous cell carcinoma (HNSCC) eligible for curative-intent resection (+/- adjuvant therapy), who receive neo-adjvuant pembrolizumab + epacadostat.

The primary objective of this study is to determine rate of major treatment effect (MTE) to neoadjuvant pembrolizumab+epacostat immunotherapy in SCCHN compared to historic data with neoadjuvant pembrolizumab alone.

DETAILED DESCRIPTION:
The KEO study is a single arm phase II trial including 44 patients with T1N1-2B, T2N0-N2B head and neck squamous cell carcinoma (HNSCC) eligible for curative-intent resection (+/- adjuvant therapy), who receive neo-adjvuant pembrolizumab + epacadostat. Patients that fit the inclusion criteria (see detailed eligibility criteria below) will receive neoadjuvant immunotherapy either with anti-PD-1 (pembrolizumab) alone or anti-PD-1 in combination with IDO1 inhibition (epacadostat). Patients will receive 200 mg IV Pembrolizumab every 3 weeks for up to 3 doses over a period of 8 weeks as well as oral epacadostat 100 mg BID starting on day 1 for the duration of pembrolizumab treatment.

All patients will undergo baseline biopsy (mandatory, sampling ≥ 4 areas to represent the tumor), as well as baseline imaging (and for exploratory analysis collection of blood for baseline ctDNA testing and TCR analysis). Patients who are unable to safely (or for other reasons unwilling to undergo biopsy at baseline and on treatment 3-4 weeks in for infiltrate assessment are not eligible for the study. MRI is the preferred imaging modality; however, diagnostic CT is acceptable if patient is unable to undergo MRI or as clinically indicated.

Subsequently at week 3-4 an interim assessment will be performed:

1. All patients will undergo imaging with a 2nd MRI scan (or CT, to match prior imaging).
2. All patients will also undergo repeat mandatory on-treatment biopsy consisting of of 4-6 representative samples to compare to the baseline biopsy. Adequacy of response to treatment will be assessed in assessing eradication of tumor/presence of antitumor tumor response (analogous to reports in lung cancer (Forde et al ESMO 2016). The on-treatment biopsy is essential in the assessment of early response and decision to extend neo-adjuvant treatment to 8 weeks is based in large part on this biopsy. In patients where an on-treatment biopsy is not obtained (e.g no longer considered safe or status of patient has changed), patients will automatically be considered non-complete responders, and take off study after 4 weeks (with the very unlikely but possible exceptions of complete response radiologic response at 4 weeks imaging).
3. For exploratory purposes, blood will also be drawn for repeat ctDNA and TCR analysis in order to assess potential suitability of dynamic changes ctDNA or TCR clonality/diversity as candidate biomarkers for follow-up studies.

At the week 3/4 interim assessment, results of the imaging and biopsy will be used to determine response and to determine continuation of immunotherapy induction treatment for up to 8 weeks (full immunotherapy induction course). Patients that demonstrate stable disease or tumor shrinkage radiographically and biopsy demonstrating dense lymphocytic infiltrate with dying tumor / decrease in residual viable tumor will continue on protocol.

Those patients with lack of lymphocytic infiltrate/dying tumor or increasing tumor on radiology (and confirmed on pathology from 2nd biopsy) will be transitioned to standard of care treatment with early salvage surgery or chemoradiation (as clinically indicated).

Pre-surgery assessment: For those patients continuing - a second confirmatory scan will be done 3-4 weeks later again coupled with a blood draw, and followed by surgery at/around week 8 (+/-1 week depending on operating schedules).

Definitive surgery will be done at week 8. Surgical specimens will again be evaluated for percentage residual viable tumor and inflammatory infiltrate. Patients that exhibit complete pathologic response (no viable tumor) will follow close observation with repeat imaging (CT/MRI at 4-6 weeks), clinical exams and a PET scan at 12 weeks post-surgery (as well as serial ctDNA draws (exploratory).

Patients with major pathologic responses (≤10% residual tumor, but tumor present) will be treated with de-escalated adjuvant radiation therapy as determined by the tumor board/radiation oncology.

Patients with a surgical specimen that demonstrates >10% residual tumor after surgery will undergo standard adjuvant RT/CRT as indicated.

Adjuvant Phase: Patients will continue adjuvant pembrolizumab plus epacadostat every 3 weeks for 12 months and be monitored with ctDNA and imaging.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Patients with non-bulky/non-bulky squamous cell carcinomas of the head and neck, with an indication for surgical therapy.

  1. T1N1-N2B, T2-4N0-N2b stage are generally eligible
  2. If determined per tumor board that a low-volume/non-bulky tumor of another stage is appropriate for resection (e.g. small volume T4 with a small amount of bone invasion) such tumors may also be considered for this study if recommendation in tumor board is such.
* Be appropriate candidates for resection and curative intent therapy in general.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Consent to undergo biopsy from a newly obtained core or excisional biopsy of a tumor lesion before study drug administration, and during treatment. Biopsy in case of progressive disease is optional.
* Ability to swallow tablets (at future point administration via G-tube may be allowed if approved by drug manufacturer)
* Measurable disease per RECIST 1.1.
* Known HPV status for oropharyngeal primary tumors.
* Pre-operative scans including MRI/CT neck and, CT chest with contrast. If contrast is contraindicated, Staging PET or PET-CT is acceptable although high quality / diagnostic cross-sectional imaging of the head and neck area is recommended.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR within upper limit of normal (ULN) OR

Measured or calculateda creatinine clearance ≥60 mL/min for subject with creatinine (GFR can also be used in place of creatinine or levels > institutional ULN CrCl)

Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN

AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN

Albumin >2.5 mg/dL

Coagulation International Normalized Ratio (INR) or ≤1.5 X ULN unless subject is receiving Prothrombin Time (PT) anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is considered an adequate contraception method.

Exclusion Criteria:

* Has a diagnosis now or in the past of immunodeficiency requiring systemic steroid therapy in excess of physiologic dose (or any other form of immunosuppressive therapy within 10 days prior to the first dose of trial treatment).
* Has bulky tumor (define as N3 lymph node or equivalent lymph conglomerate (≥ 6 cm in one dimension), or primary tumor > 4 cm). Cystic HPV+ lymph nodes should be assessed in tumor board and may not be considered bulky.
* Has a known history of active TB (Bacillus Tuberculosis).
* Other life-threatening illness that is expected to impact life expectancy within 3 years.
* Hypersensitivity to pembrolizumab, epacadostat or any of its excipients.
* Has a known additional malignancy that was diagnosed within the last five years that is either progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, or in a broader sense is not felt to impact life-expectancy.
* Has active autoimmune disease that has required systemic (large physiologic dose) treatment in the past year (i.e. with use of disease modifying agents, corticosteroids or any other immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic immunosuppressive treatment.
* History of non-infectious pneumonitis requiring steroids or current pneumonitis
* Has an active viral infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Allogeneic organ or stem cell transplant
* History of interstitial lung disease (ILD)/pneumonitis requiring treatment with steroids and patients with active ILD/pneumonitis

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Rate of major treatment effect (rate of treatment response) | 3-4 weeks after patient has begun treatment
  MTE will be assessed in the same way as done by Uppaluri et al (Uppaluri ASCO 2017) upon pathologic review and assessment of 50% resolution of tumor with active immune response (termed "major treatment effect" in their study).
Rate of complete response | 8 weeks after patient has begun treatment
  Response rate at surgery compared to historic data with chemotherapy

SECONDARY OUTCOMES:
Progression free survival rate | From the start of treatment to the first documented report of disease progression or death, whichever comes first, not to exceed 100 months.
Overall survival rate | From the start of treatment to the time of death, not to exceed 100 months.
Number of patients with adverse events prior to and after surgery | Up to 2 years
Complete response rate | From the start of treatment to the first documented report of response, disease progression, or death, whichever comes first, not to exceed 100 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States